**ID:** 130852.

Study: COVID-19: Healthcare Worker

Bioresource: Immune Protection and

Pathogenesis in SARS-CoV-2.

NCT Number: 04318314.

Document Date: Updated on 01/05/2021.

**Title of document:** List of current published, in press, preprints and under review articles written from the study.

## Published/In press:

- 1. <u>www.covidsortium.com</u> Website.
- 2. <u>Wellcome open:</u> Study design.
- 3. PLOS1: academic research impact of COVID-19
- 4. <u>Lancet:</u> Serial falling PCR levels in Healthcare Workers
- 5. Circulation: Myocardial injury from COVID-19.
- 6. <u>Lancet:</u> follow-up PCR positivity levels in in Healthcare Workers
- 7. <u>Science Immunology:</u> T cell, serology and neutralising antibody heterogeneity in mild disease.
- 8. <u>European Heart Journal</u>: Patterns of myocardial injury from COVID-19.
- 9. Lancet E-BioMed: Antibody dynamics in mild SARS-CoV-2 infection.
- 10. JACC Imaging: Cardiovascular late effects of mild disease.
- 11. <u>Lancet:</u> Second booster vaccine not necessary after prior COVID-19.
- 12. <u>E-ClinMed:</u> Infection risk, BAME and health role.
- 13. <u>Science</u>: Impact of vaccination on T and B cell response to variants: (in press, fast track).

## Preprints/under review

- 14. Viral transcriptomics paper: Under review Lancet microbe.
- 15. Whole genome transcriptomics signature mild disease.